CLINICAL TRIAL: NCT02499965
Title: The Use of a Topical Anesthetic Skin Refrigerant to Reduce the Pain Associated With Intravenous Catheter Insertion, A Double Blinded, Patient/Placebo Controlled, Study
Brief Title: Skin Refrigerant to Reduce the Pain Associated With IV Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kurt Fossum, Major, USA, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 404187-2
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Pain
Keywords: Topical Anesthetic; Ethyl Chloride; Pain Reduction; IV cannulation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical Ethyl Chloride (Product B) (Active Comparator): Ethyl Chloride Topical Aerosol Anesthetic applied to arm
  Interventions: Drug: Ethyl Chloride Topical Aerosol Anesthetic
- Topical Sterile Water (Product A) (Placebo Comparator): Nature's Tears Sterile water in an aerosol can
  Interventions: Drug: Nature's Tears Sterile Water

INTERVENTIONS:
Drug: Ethyl Chloride Topical Aerosol Anesthetic — Sprayed on the skin for 5-8 seconds immediately before IV cannulation
  Other Names: Study Device or Product B
  Arms: Topical Ethyl Chloride (Product B)
Drug: Nature's Tears Sterile Water — Sprayed on the skin for 5-8 seconds immediately before IV cannulation
  Other Names: Placebo or Product A
  Arms: Topical Sterile Water (Product A)

SUMMARY:
The purpose of this study is to determine whether or not the pain of IV catheter insertion in the Emergency Department can be reduced significantly with the use of a rapid acting topical anesthetic spray and to determine whether or not healthcare providers who undergo such treatment are likely to endorse its use in their future practice.

DETAILED DESCRIPTION:
We recruited 38 emergency department healthcare providers (doctors, physician assistants, nurses and medics) to receive a total of two separate IV canulations - one in one arm and the other in the other. One IV canulation would be pretreated with Ethyl Chloride topical anesthetic (the study product) and the other would be pre-treated with a placebo (sterile water in an aerosol can). Both the participants and the nurses, PAs and medics who placed the IVs were blinded as to which was the Ethyl Chloride and which was the placebo. After the IVs were placed the participants were asked to rate the pain of IV canulation on a scale of 1 to 10 for each of the pre-treatments, to state which one they believed to be superior in reducing the pain of receiving the IV, to state whether or not they would like the intervention that they rated as superior to be used on themselves and finally how likely they were on a 5 point scale to incorporate the intervention they rated as superior into their future practice.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. A healthcare worker who routinely orders or places IV catheters.
3. Consents to participate in the study.

Exclusion Criteria:

1. History of hypersensitivity to Ethyl Chloride.
2. Break, or swollen in the skin at the proposed IV site.
3. Pregnancy or lactating female.
4. Recent tattoo in either of the two proposed anatomical areas for IV cannulation.
5. Skin infection in either of the two proposed anatomical areas for IV cannulation.
6. Missing a contralateral limb to place the second IV.
7. Recent trauma to one of the upper extremities or any neuropathic or radicular condition that could affect the participant's perception of pain in the antecubital fossa of each arm.

   -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pain | 1 minute
  Ordinal pain scale (1-10)

SECONDARY OUTCOMES:
Preferred product | 1 minute
  Categorical selection of preferred product for use on self prior to IV placement
Desire to use on self in future | 1 minute
  Binary (yes, no) desire to use on self prior to IV placement in future
Desire to use on patients in future | 1 minute
  Binary (yes, no) desire to use on patients prior to IV placement in future
Likelihood to use on patients in future | 1 minute
  5 point likert scale ranging from "very unlikely" to "very likely"

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Fossum, MPAS, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Fung S, Phadke CP, Kam A, Ismail F, Boulias C. Effect of topical anesthetics on needle insertion pain during botulinum toxin type A injections for limb spasticity. Arch Phys Med Rehabil. 2012 Sep;93(9):1643-7. doi: 10.1016/j.apmr.2012.03.012. Epub 2012 Mar 23. PMID 22449552
- [Background] Mawhorter S, Daugherty L, Ford A, Hughes R, Metzger D, Easley K. Topical vapocoolant quickly and effectively reduces vaccine-associated pain: results of a randomized, single-blinded, placebo-controlled study. J Travel Med. 2004 Sep-Oct;11(5):267-72. doi: 10.2310/7060.2004.19101. PMID 15544709
- [Background] Hartstein BH, Barry JD. Mitigation of pain during intravenous catheter placement using a topical skin coolant in the emergency department. Emerg Med J. 2008 May;25(5):257-61. doi: 10.1136/emj.2006.044776. PMID 18434455
- [Background] Farion KJ, Splinter KL, Newhook K, Gaboury I, Splinter WM. The effect of vapocoolant spray on pain due to intravenous cannulation in children: a randomized controlled trial. CMAJ. 2008 Jul 1;179(1):31-6. doi: 10.1503/cmaj.070874. PMID 18591524
- [Background] Hijazi R, Taylor D, Richardson J. Effect of topical alkane vapocoolant spray on pain with intravenous cannulation in patients in emergency departments: randomised double blind placebo controlled trial. BMJ. 2009 Feb 10;338:b215. doi: 10.1136/bmj.b215. PMID 19208703
- [Background] Costello M, Ramundo M, Christopher NC, Powell KR. Ethyl vinyl chloride vapocoolant spray fails to decrease pain associated with intravenous cannulation in children. Clin Pediatr (Phila). 2006 Sep;45(7):628-32. doi: 10.1177/0009922806291013. PMID 16928840
- [Background] Ducharme, J. (2011). Acute Pain Management in Adults. In J. E. Tintinalli, J. S. Stapczynski, O. J. Ma, D. M. Cline, R. K. Cydulka, & G. D. Meckler, Tintinalli
- [Derived] Fossum K, Love SL, April MD. Topical ethyl chloride to reduce pain associated with venous catheterization: a randomized crossover trial. Am J Emerg Med. 2016 May;34(5):845-50. doi: 10.1016/j.ajem.2016.01.039. Epub 2016 Feb 13. PMID 26971823